CLINICAL TRIAL: NCT02725801
Title: Randomized Clinical Trial Comparing 1-Port and 2-Port Tissue Expanders for Breast Reconstruction
Brief Title: Comparison of One-port and Two-port Tissue Expanders for Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesley Wong (Other)
Responsible Party: Sponsor-Investigator, Lesley Wong, Associate Professor of Plastic Surgery, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-0064
Record Dates: First submitted 2016-02-27; First posted 2016-04-01 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- one-port (Active Comparator): intervention is placement of one-port tissue expander at time of reconstruction
  Interventions: Device: Allergen one-port tissue expander placement
- two-port (Active Comparator): intervention is placement of two-port tissue expander at time of reconstruction
  Interventions: Device: AlloX2 two-port tissue expander placement

INTERVENTIONS:
Device: Allergen one-port tissue expander placement — patients will be randomized to receive a one port or two port tissue expander for breast reconstruction
  Other Names: Allergen one-port tissue expander
  Arms: one-port
Device: AlloX2 two-port tissue expander placement — patients will be randomized to receive a one port or two port tissue expander for breast reconstruction
  Other Names: AlloX2 two-port tissue expander
  Arms: two-port

SUMMARY:
Appropriate patients undergoing going immediate breast reconstruction with tissue expanders following mastectomy will be randomized to receive one-port or two-ports tissue expanders. Their clinical course, complications, and outcome will be analyzed.

DETAILED DESCRIPTION:
The goal of this study is to compare a traditional single port expander with a two-port expander for equivalency when used for breast reconstruction following mastectomy. Complication rates that will be tracked include seroma, mastectomy skin flap necrosis, infection, wound dehiscence, need for explantation of the expander. Management of seromas will be compared between the two groups. The investigators hypothesize that the AlloX2 expander will be as effective in achieving the final outcome of completion of the second stage of reconstruction with equal or improved complication rates.

Study Design A prospective 1:1 randomized, single center, open label study will compare the traditional 1- port tissue expander with the AlloX2 2-port expander placed during immediate tissue expander breast reconstruction. Due to the nature of the surgery, the study cannot be blinded. Patients will be followed until completion of expansion and exchange for the permanent implant which typically takes 2 to 3 months. Risks factors that have been previously identified to be associated with increased postoperative complications include smoking, obesity, breast size, diabetes, radiation therapy, and expander fill volume will be identified. The final outcome is completion of expansion and exchange to permanent implant.

Standard operative procedure and postoperative care will be done. Both groups will have the same two external drains placed which is standard operative procedure. Complications will be noted at each postoperative clinic visit and entered into a database. Complication rates will be compared between the two groups and associations with risk factors will be analyzed. There will be no cross-over into the other group in case of reconstructive failure. Treatment failures will be treated in the same fashion in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patient agrees to immediate tissue expander breast reconstruction
* a suitable patient for tissue expander reconstruction

Exclusion Criteria:

* not a surgical candidate for immediate breast reconstruction
* age less than 18
* patient declines tissue expander reconstruction
* patient anticipated to need radiation therapy postoperatively

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2019-07-19 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Wong, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One-port | Two-port
Started | 8 | 12
Completed | 8 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One-port | Two-port | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.75 (12.28) | 51.08 (13.83) | 48.92 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Replacement of Tissue Expander With Permanent Implant
Description: The number of patients that are able to undergo replacement of the tissue expander between the two arms will be compared
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | One-port | Two-port
Number analyzed (Participants) | 8 | 12
Participants | 8 | 12

2. Secondary Outcome: Number of Participants Who Required Additional Intervention
Description: Number of participants requiring additional intervention following tissue expander placement will be compared between the two arms of the study
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | One-port | Two-port
Number analyzed (Participants) | 8 | 12
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: 3 months
Description: All-cause mortality was not monitored/assessed.
Arm/Group | One-port | Two-port
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/8 | 4/12
Other Adverse Events (participants affected / at risk) | 0/8 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One-port (N=8) | Two-port (N=12)
re-operation (Surgical and medical procedures) | 1 (1) | 4 (4) — Reoperation for infection or seroma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT02725801/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT02725801/ICF_001.pdf